CLINICAL TRIAL: NCT04546217
Title: Gait Training Combined With Strategies to Induce Transference to Real Life for People With Stroke
Brief Title: Gait Training Combined With Behavioral Strategies for People With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Sarah dos Anjos, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300005407
Record Dates: First submitted 2020-08-25; First posted 2020-09-11 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Gait, Hemiplegic; Behavior and Behavior Mechanisms
Keywords: Gait training; Robotic training; Transference; Behavioral strategies
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will not be involved nor present during the training sessions. Also the outcome assessments will be performed without the presence of the interventionist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treadmill training +Transfer package (TT+TP) (Experimental): The TT+TP group will receive 24 sessions (3x week for 8 weeks) of robotic treadmill gait training in a robotic device called KineAssist. In combination with the gait training, participants in this group will also receive a group of behavioral strategies called the "Transfer Package" (TP). Each intervention session will last 1.5h, 1h for the gait training and 30 minutes dedicated for the transfer package.
  Participants will be assessed pre-, post-intervention, 3 and 6 months after the end of the intervention. Also, participants will be interviewed to investigate their perceptions about each element of the intervention, benefits, side effects and suggestion for change.
  Interventions: Combination Product: Treadmill training + transfer package (TT+TP)
- Treadmill training (TT) (Active Comparator): The TT group will receive 24 sessions (3x week for 8 weeks) of robotic treadmill gait training in a robotic device called KineAssist.
  Participants will be assessed pre-, post-intervention, 3 and 6 months after the end of the intervention. Also, participants will be interviewed to investigate their perceptions about each element of the intervention, benefits, side effects and suggestion for change.
  Interventions: Device: Treadmill training (TT)

INTERVENTIONS:
Combination Product: Treadmill training + transfer package (TT+TP) — Participants will walk in different speeds, step over obstacles, and keep their balance during perturbations in the robotic treadmill. In combination with the gait training, participants will also receive a group of behavioral strategies (Transfer Package). Participants will sign the behavioral contract to achieve safety while engaging in activities, increase use of the paretic leg in daily activities, and increase coordination of both legs. A list of activities to be performed outside the clinical setting, the Home Skill Assignment, will be developed for each day of the week during the treatment period and given to the participants at the end of the session. The Home Practice after treatment aims to assure continued progress with LE use after the intervention program is completed. The LE-MAL Log will be administered in all sessions to assess quality of movement of the affected leg, level of assistance needed to perform daily activities, and level of confidence.
  Arms: Treadmill training +Transfer package (TT+TP)
Device: Treadmill training (TT) — Participants in this group will walk in different speeds, step over obstacles, and keep their balance during perturbations in the robotic treadmill. The treadmill training will be identical to the experimental group, but no element of the TP will be delivered.
  Arms: Treadmill training (TT)

SUMMARY:
A variety of rehabilitation techniques focused on improving disability after stroke have shown significant changes on walking speed, and endurance. Also, the administration of combined techniques showed better results. Previous studies have suggested that embedding behavioral strategies in neurorehabilitation protocols can enhance patient's adherence and participation outside the clinical setting. The addition of a group of behavioral strategies called Transfer Package (TP) has been widely used in motor training protocol (e.g. Constraint-Induced Movement Therapy). The TP has shown to enhance the effects of treatment 2.4 times when compared to motor training alone. However, the effect of TP when combined with robotic gait training remains unexplored. In this study our goal is to combine the TP with robotic gait training. The hypothesis is that using the TP in combination with robotic gait training will enhance the outcome of robotic gait training alone and will induce long term transference and retention of the motor skills observed after treatment. More importantly, this experimental intervention is more meaningful to the patient and can be more easily implemented on the clinical setting. The aims of this study are (1) to assess transfer and long-term retention of walking and balance skills after robotic treadmill gait training combined with the TP, (2) to understand participants' acceptability and perceptions of the TP as a tool to enhance transfer of skills to real-world situations, and (3) to examine the feasibility of these combined intervention to improve walking and balance after stroke.

DETAILED DESCRIPTION:
This proposal seeks to investigate the effect of gait training combined with behavioral strategies on long-term retention of improvements on gait parameters and use of the affected lower-extremity in real-world situations.

Aim 1: To assess transfer and long-term retention of walking and balance skills after robotic treadmill gait training combined with the TP. A total of 24 participants with chronic stoke will be randomly allocated to either treadmill training combined with the TP (TT+TP) or usual TT with an educational approach. The 8-week intervention will consist of three weekly sessions of 1 hour of TT. The experimental group will also receive the TP for 30 minutes and the control group will receive a manual with exercises to be performed at home. The primary outcome is the change in Lower-Extremity Motor Activity Log. Also, change in walking speed, endurance, functional strength and use of the affected LE will be assessed at 3- and 6-months after the intervention.

Aim 2: To understand participants' acceptability and perceptions of the TP as a tool to enhance transfer of skills to real-world situations. A qualitative approach will be used for evaluating the acceptability of the TT + TP protocol. Individual interviews will be conducted with all participants to assess their opinion about TP, particularly, their perceived influence of the TP on real-life situations.

Aim 3: To examine the feasibility of body weight support treadmill training combined with behavioral strategies to improve walking and balance after stroke. Compliance with the intervention will be measured as the number of sessions attended and number of activities performed outside the clinical setting. Also, the relationship between the outcome changes after the intervention and the participants' perceptions will be explored.

The hypothesis is that the use of the TP will promote long-term retention of the positive changes in walking and balance and also changes in real-world situations. This pilot study will lead to future studies with larger samples in order to compare the effect of body weight support treadmill training combined with the TP. The long-term goal is to provide a systematic combination of strategies to improve gait and mobility after stroke that can be implemented in the clinical setting.

In this study our goal is to combine gait training with a robotic treadmill and the TP. The TP is adapted from our previous work with Lower-Extremity Constraint-Induced Movement Therapy. The effect of the combined gait training will on real-world use of the affected lower extremity, walking speed, endurance, functional strength will be tested as well as the effect of the TP on long-term retention. Furthermore the combined TP + treadmill training will be meaningful to the patient.

1. Participants: sampling and selection criteria Participants will be recruited from a list of patients that have been discharged from the Spain Rehabilitation Center at University of Alabama at Birmingham (UAB). Participants will be recruited from a registry of individuals who have had a stroke and whom are interested in research managed by the Department of Neurology at UAB.

   The inclusion criteria is as follows: (1) 18 years of age or older; (2) at least 6 months post stroke; (3) present lower extremity motor impairment secondary to stroke, (4) able to walk at least 10 feet with or without personal assistance; (5) discharged from rehabilitation. Participants will be excluded if present uncontrolled clinical conditions, weight > 400lb because this is limit supported by the KineAssist, other neurologic conditions, a Mini-Mental State Examination score (MMSE) <24, inability to provide the informed consent, and insufficient language skills to answer the screening, assessments and interview questions.

   Participants will be first contacted by phone and the study will be fully explained, if the participant is interested the first screening interview will be conducted. During this first screening the inclusion criteria and the availability of the participants will be checked. After assuring the inclusion criteria have been met, a more thorough in-person screening examination will be scheduled in order to assess participants' cognitive and motor functions. All participants will be asked to voluntarily provide informed consent.

   A total of 24 people with chronic stroke will be selected and will be randomly allocated to TT+TP (N=12) or TT group (N=12). Sample calculation was performed using standard deviation and effect size of the LE-MAL which was obtained from a previous study conducted by the PI.20 This proposal is 90.9% powered to detect a significant difference between study arms of 1.55 improvement on the LE-MAL.
2. Intervention All participants will receive the same robotic treadmill training. The training conducted on the robotic treadmill device will be based on different constructs of walking and balance, including standing, stepping, propulsion, speed, strength, and endurance. The KineAssistTM (KA) robotic device will be used for targeted training of participants. The KA uses a patented force-sensing, pelvic support mechanism to sense the user's intended walking speed and direction to drive a moving surface, thus allowing a person to move at their own intended walking speed and pace. The device is sensitive enough to allow sudden starting and stopping movements, so that balance tasks and responses to sudden disturbances can be accommodated. This system is uniquely different compared to a treadmill, which only moves at a fixed speed and can only allow repetitive stepping protocols. The robotic system that allows individuals to move at self-driven speeds against challenging conditions in order to implement a combinatorial approach to assessment and intervention.

   The transfer package element of the body weight support treadmill training, was modified accordingly in order to fit the gait training intervention. The TP procedures will be administered as described below.

   On the first day of treatment, participants will be asked to sign the behavioral contract (BC). The purpose of the BC is to: (1) achieve safety while engaging in improved use of the LEs, (2) increase use of the more-affected LEs in functional activities whenever possible, and (3) increase use of both LEs in a more coordinated manner. Additionally, the behavioral contract formally engages the patient in actively exploring more ways to use their more-affected LE in their home environment and in adopting a problem-solving approach to accomplish that end. The BC will be worked out with the patient at the end of the first treatment day. Before discussing the contract, therapist will develop in conjunction with the participant a daily activity schedule from the time of awakening in the morning until arrival at the clinic for training on subsequent days, and between sessions..

   Also a list of activities to be performed outside the clinical setting, the Home Skill Assignment (HSA), will be developed for each day of the week during the treatment period. The HSA process is a transfer technique designed to encourage use of the more-affected LE during activities of daily living (ADL). The HSA supports and should be in agreement with the behavioral contract. It will be given to the patient as a written set of activities to be accomplished after the end of the treatment session and it has a check-off component. After each activity is accomplished outside the treatment setting the patient checks that item Another component of the TP is the Home Practice after treatment. The purpose of home task practice after the intervention period is to assure continued progress with LE use after the intervention program is completed. With home practice, participants are encouraged to engage in functional skills and fitness activities on a daily basis. These activities will maintain improvements in LE use realized during the LE-CIMT protocol and possibly enhance them. Toward the end of treatment, a written individualized post-treatment home practice program will be developed and given to the patient. The program consists of 7 separate lists, one for each day of the week, repeated weekly.

   The last TP element is the administration of the Lower-Extremity Motor Activity Log (LE-MAL) during all treatment sessions. A full description of the LE-MAL is provided in the Results/Outcomes section below.

   The 8-week intervention will consist of three weekly sessions of 1 hour of TT. The experimental group will also receive the TP for 30 minutes and the control group (TT group) will receive a handbook with exercises and stretching techniques. Therapists will ask the participants of this group to pick up at least 2-3 activities and perform them for 30 minutes everyday.
3. Outcomes In order to assess LE physical performance and use, the following primary outcome tools will be used: (1) the primary outcome is the Lower Extremity Motor Activity Log (LE-MAL);20,21 (2) Berg Balance Scale (BBS);22 (3) 10 meters walk test (10MWT);23 and (4) 6 minutes walking test (6MWT).24 The secondary outcomes are: (1) 5 times sit to stand (5TSTS);25 (2) Fear of Falling Avoidance Behavior Questionnaire (FFABQ).36 The LE-MAL is a semi-structured interview, created in the UAB Constraint-Induced Therapy Research Group laboratory, that consists of questions asking the participant the level of assistance, how well her/his performance is, and level of confidence while executing 14 different daily tasks (e.g. walking indoors, climbing stairs) in real world environment.20,41 The LE-MAL investigates the transference of the skills addressed during the treatment to different contexts. The principal investigator of this proposal has used the test extensively and has participated in a reliability and validity study of the LE-MAL which showed that the LE-MAL is a reliable tool in both test-retest results (r=0.93) and internal consistency (Cronbach's alpha = 0.96).

Assessments will be administered during pre-, post-treatment and follow up visits (3 and 6 months after the end of the intervention protocol). Each assessment visit will last approximately 40 minutes. The follow up assessment will provide information regarding long-term retention of results and will serve as the basis for future research. Pre-, post-treatment, and follow up assessments will be compared in order to investigate changes observed compared to the baseline and long term retention of these changes. For this, an analysis of covariance (ANCOVA) will be utilized to analyze the changes among different time points (post-treatment and follow up assessments). Those subjects with complete data will contribute to the analysis. In case of missing data, a last observation carried forward (LOCF) sensitivity analysis will be conducted. In addition, those with incomplete follow-up data will be compared to subjects with complete data to see if the groups differ significantly in baseline characteristics.

Compliance will be described by the percentage of sessions attended and number of activities performed outside the clinical setting. Considering that the participants will receive a list with 10 activities to be performed in the real world (Home Skill assignment), a total of 560 activities will be listed during the intervention. In a previous LE Constraint-induced therapy study, participants performed approximately 85% of the activities. However, this was a shorter intervention (2 weeks) and a lower percentage might be observed in longer protocol as the purposed here. Thus, a minimum of 60% of compliance regarding the list of activities will be expected.

A qualitative strand will be conducted after the conclusion of the treatment. Participants will be interviewed face-to-face to determine perspectives regarding the intervention protocol, especially acceptability. Semi-structured, in-depth interviews will be conducted regarding how time consuming the TP is (outside the clinical setting), potential routine modifications, and potential suggestions. The interviews will be conducted by other researchers who are knowledgeable and skilled in qualitative interviewing and are uninvolved in the delivery of the treatment to avoid influence on participants' responses. The interviews will be audio recorded and transcribed verbatim. The interviewer will follow a script which provides participants with an overview of the interview protocol. The interview questions will include participant's impression about the elements of the TP, the transference of motor skills trained during the gait sessions to other environments, compliance with procedures, and suggestions for modifications. Perceptions regarding the control condition will also be collected using the same procedures.

The qualitative data will be analyzed through thematic analysis procedures in which the main themes collected along the interview will be categorized and reported.27 Two researchers will code the transcripts independently. The themes will be compared and revised by both coders. The themes will be refined if needed, and the final list of themes will be reported in a joint display.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* at least 6 months post stroke;
* present lower extremity motor impairment secondary to stroke;
* able to walk at least 10 feet with or without personal assistance;
* discharged from rehabilitation.

Exclusion Criteria:

* presence of uncontrolled clinical conditions;
* weight > 400lb because this is limit supported by the KineAssist
* other neurologic conditions;
* Mini-Mental State Examination score (MMSE) <24;
* inability to provide the informed consent;
* insufficient language skills to answer the screening, assessments and interview questions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehrholz J, Thomas S, Elsner B. Treadmill training and body weight support for walking after stroke. Cochrane Database Syst Rev. 2017 Aug 17;8(8):CD002840. doi: 10.1002/14651858.CD002840.pub4. PMID 28815562
- [Background] Taub E. Harnessing brain plasticity through behavioral techniques to produce new treatments in neurorehabilitation. Am Psychol. 2004 Nov;59(8):692-704. doi: 10.1037/0003-066X.59.8.692. No abstract available. PMID 15554826
- [Background] Taub E, Uswatte G, Mark VW, Morris DM, Barman J, Bowman MH, Bryson C, Delgado A, Bishop-McKay S. Method for enhancing real-world use of a more affected arm in chronic stroke: transfer package of constraint-induced movement therapy. Stroke. 2013 May;44(5):1383-8. doi: 10.1161/STROKEAHA.111.000559. Epub 2013 Mar 21. PMID 23520237
- [Background] Morris DM, Taub E, Mark VW. Constraint-induced movement therapy: characterizing the intervention protocol. Eura Medicophys. 2006 Sep;42(3):257-68. PMID 17039224
- [Background] Mark VW, Taub E. Constraint-induced movement therapy for chronic stroke hemiparesis and other disabilities. Restor Neurol Neurosci. 2004;22(3-5):317-36. PMID 15502259
- [Background] Stretton CM, Mudge S, Kayes NM, McPherson KM. Interventions to improve real-world walking after stroke: a systematic review and meta-analysis. Clin Rehabil. 2017 Mar;31(3):310-318. doi: 10.1177/0269215516640863. Epub 2016 Jul 10. PMID 27056251
- [Background] Mark VW, Taub E, Uswatte G, Bashir K, Cutter GR, Bryson CC, Bishop-McKay S, Bowman MH. Constraint-induced movement therapy for the lower extremities in multiple sclerosis: case series with 4-year follow-up. Arch Phys Med Rehabil. 2013 Apr;94(4):753-60. doi: 10.1016/j.apmr.2012.09.032. Epub 2012 Oct 27. PMID 23111280
- [Background] Dos Anjos SM, Morris DM, Taub E. Constraint-Induced Movement Therapy for Improving Motor Function of the Paretic Lower Extremity After Stroke. Am J Phys Med Rehabil. 2020 Jun;99(6):e75-e78. doi: 10.1097/PHM.0000000000001249. PMID 31246610
- [Background] Dos Anjos S, Morris D, Taub E. Constraint-Induced Movement Therapy for Lower Extremity Function: Describing the LE-CIMT Protocol. Phys Ther. 2020 Apr 17;100(4):698-707. doi: 10.1093/ptj/pzz191. PMID 31899495
- [Background] Berg K, Wood-Dauphinee S, Williams JI. The Balance Scale: reliability assessment with elderly residents and patients with an acute stroke. Scand J Rehabil Med. 1995 Mar;27(1):27-36. PMID 7792547
- [Background] Green J, Forster A, Young J. Reliability of gait speed measured by a timed walking test in patients one year after stroke. Clin Rehabil. 2002 May;16(3):306-14. doi: 10.1191/0269215502cr495oa. PMID 12017517
- [Background] Eng JJ, Dawson AS, Chu KS. Submaximal exercise in persons with stroke: test-retest reliability and concurrent validity with maximal oxygen consumption. Arch Phys Med Rehabil. 2004 Jan;85(1):113-8. doi: 10.1016/s0003-9993(03)00436-2. PMID 14970978
- [Background] Mong Y, Teo TW, Ng SS. 5-repetition sit-to-stand test in subjects with chronic stroke: reliability and validity. Arch Phys Med Rehabil. 2010 Mar;91(3):407-13. doi: 10.1016/j.apmr.2009.10.030. PMID 20298832
- [Background] Landers MR, Durand C, Powell DS, Dibble LE, Young DL. Development of a scale to assess avoidance behavior due to a fear of falling: the Fear of Falling Avoidance Behavior Questionnaire. Phys Ther. 2011 Aug;91(8):1253-65. doi: 10.2522/ptj.20100304. Epub 2011 Jun 23. PMID 21700763
- [Result] Pollock A, Baer G, Campbell P, Choo PL, Forster A, Morris J, Pomeroy VM, Langhorne P. Physical rehabilitation approaches for the recovery of function and mobility following stroke. Cochrane Database Syst Rev. 2014 Apr 22;2014(4):CD001920. doi: 10.1002/14651858.CD001920.pub3. PMID 24756870

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was delayed due to the SARS-COVID pandemic. Thus, instead of the initial 24 participants, a 2:1 ratio was used targeting to enroll at least 18 individuals. This way, from the total 19 individuals included in this study, 12 were assigned to the TT+TP and 7 to the TT.
  Participants were recruited from a list of patients from the Spain Rehabilitation Center at UAB or were referred by UAB physicians and therapists.
  Recruitment were conducted from October 2020 to April 2022.
Pre-assignment Details: The of the study started during the SARS-COVID pandemic, leading to challenges on recruitment, scheduling due to institutional and individual restrictions. Considering that the study participants were considered at high risk to develop severe symptoms if contracted the virus, the first participant started 8 months after was predicted, and the number of participants needed to be reduced to accommodate institutional restrictions and follow the timeline provided by the funding source.
Groups:
- Treadmill Training +Transfer Package (TT+TP): The TT+TP group received 18 1.5h sessions (3x for 6 weeks) of robotic treadmill (KineAssist) gait training. In combination with the gait training, participants in this group received the "Transfer Package" (TP). On each session, 1h was allocated for the gait training and 30 minutes for the TP. As part of the TP, participants signed a behavioral contract to achieve safety while engaging in activities outside the clinic, increase use of their paretic leg in daily activities, and increase coordination of both legs. The TP also included a list of activities to be performed outside the clinical setting, the Home Skill Assignment, that was developed daily during the treatment period and given to the participants at the end of the session. There were also the Home Practice after treatment to assure continued progress with LE use after the intervention program is completed. The Lower Extremity Motor Activity Log (LE-MAL) was administered in all sessions to assess quality of movement of the affected leg, level of assistance needed to perform daily activities, and level of of confidence that their are able to maintain their balance during activity performance.
  Participants were assessed pre-, post-intervention, 3 and 6 months after the end of the intervention. Also, participants will be interviewed to investigate their perceptions about each element of the intervention, benefits, side effects and suggestion for change.
  confidence.
- Treadmill Training (TT): The TT group will receive 18 sessions (3x week for 6 weeks) of robotic treadmill gait training in a robotic device called KineAssist.
  Participants will be assessed pre-, post-intervention, 3 and 6 months after the end of the intervention. Also, participants will be interviewed to investigate their perceptions about each element of the intervention, benefits, side effects and suggestion for change.
  Treadmill training (TT): Participants in this group will walk in different speeds, step over obstacles, and keep their balance during perturbations in the robotic treadmill. The treadmill training will be identical to the experimental group, but no element of the TP will be delivered.
Period: Overall Study
Arm/Group | Treadmill Training +Transfer Package (TT+TP) | Treadmill Training (TT)
Started (Training sessions.) | 12 | 7
Completed | 9 | 7
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Uncontrolled hypertension | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treadmill Training +Transfer Package (TT+TP): The TT+TP group will receive 24 sessions (3x week for 8 weeks) of robotic treadmill gait training in a robotic device called KineAssist. In combination with the gait training, participants in this group will also receive a group of behavioral strategies called the "Transfer Package" (TP). Each intervention session will last 1.5h, 1h for the gait training and 30 minutes dedicated for the transfer package.
  Treadmill training + transfer package (TT+TP): Participants will walk in different speeds, step over obstacles, and keep their balance during perturbations in the robotic treadmill. In combination with the gait training, participants will also receive a group of behavioral strategies (Transfer Package). Participants will sign the behavioral contract to achieve safety while engaging in activities, increase use of the paretic leg in daily activities, and increase coordination of both legs. A list of activities to be performed outside the clinical setting, the Home Skill Assignment, will be developed for each day of the week during the treatment period and given to the participants at the end of the session. The Home Practice after treatment aims to assure continued progress with LE use after the intervention program is completed. The LE-MAL Log will be administered in all sessions to assess quality of movement of the affected leg, level of assistance needed to perform daily activities, and level of confidence.
- Treadmill Training (TT): The TT group will receive 24 sessions (3x week for 8 weeks) of robotic treadmill gait training in a robotic device called KineAssist.
  Participants will be assessed pre-, post-intervention, 3 and 6 months after the end of the intervention. Also, participants will be interviewed to investigate their perceptions about each element of the intervention, benefits, side effects and suggestion for change.
  Treadmill training (TT): Participants in this group will walk in different speeds, step over obstacles, and keep their balance during perturbations in the robotic treadmill. The treadmill training will be identical to the experimental group, but no element of the TP will be delivered.
- Total: Total of all reporting groups
Arm/Group | Treadmill Training +Transfer Package (TT+TP) | Treadmill Training (TT) | Total
Number analyzed (Participants) | 12 | 7 | 19
Age, Continuous [Mean (Full Range); unit: years] | 50 [42 to 63] | 53.1 [34 to 73] | 51.2 [34 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 11 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 7 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 2 | 10
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 7 | 19
NeuroQOL - Quality of Life in Neurological Disorders [Mean (Standard Deviation); unit: units on a scale] — The NeuroQOL is a self-report quality of life measure. For this study, only the Lower Extremity Function/Mobility scale was administered. The total score of the Lower Extremity Function/Mobility scale of the NeuroQOL ranges from 8-40, including 8 activities that are scores from 1-5 where 1 denotes inability to perform daily activities, and 5 no difficult in performing these tasks.
  units on a scale | 28 (5.6) | 26.9 (4.5) | 27.6 (5.3)
Time since stroke [Mean (Full Range); unit: years] | 2.0 [0.9 to 4.3] | 2.6 [0.6 to 10.2] | 2.2 [0.6 to 10.2]
Affected side [Count of Participants; unit: Participants]
  Left side | 4 | 4 | 8
  Right side | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Lower Extremity Motor Activity Log - Real World Use of the Affected Lower Extremity in Daily Activities.
Description: It is a semi-structured interview that consists of questions asking the participant the level of assistance, how well her/his performance is, and level of confidence while executing 14 different daily tasks (e.g. walking indoors, climbing stairs) in real world environment. The LE-MAL investigates the transference of the skills addressed during the treatment to different contexts. The LE-MAL is a reliable tool in both test-retest results (r=0.93) and internal consistency (Cronbach's alpha = 0.96). The score range from 0-10, where 0 is a higher level of assistance, worse quality and movement and less confidence, and 10 is given when no assistance is needed, good quality of movement is reported and the person feels completely confident in performing the activity without falling.
Time Frame: Pre-treatment (baseline), post-treatment (immediately after the last training session, at the end of week 6 of intervention), 3 months follow up post-intervention, and 6 months follow up post-intervention.
Population: COVID affected the duration of the program, which changed from 8 to 6 weeks. Overall, 5 out of 19 individuals were excluded or withdrawn. From those, 1 from the TT group completed the training sessions, but could not progress on the training, receiving 18 sessions of only endurance training instead of 6 sessions of each endurance, strengthening, and speed training. From the TT+TP group, 4 were exclude: 1 for transportation issues, 2 were not available, and 1 due to uncontrolled hypertension.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Treadmill Training +Transfer Package (TT+TP): The TT+TP group will receive 24 sessions (3x week for 8 weeks) of robotic treadmill gait training in a robotic device called KineAssist. In combination with the gait training, participants in this group will also receive a group of behavioral strategies called the "Transfer Package" (TP). Each intervention session will last 1.5h, 1h for the gait training and 30 minutes dedicated for the TP. As part of the TP, participants will sign the behavioral contract to achieve safety while engaging in activities, increase use of the paretic leg in daily activities, and increase coordination of both legs. A list of activities to be performed outside the clinical setting, the Home Skill Assignment, will be developed for each day of the week during the treatment period and given to the participants at the end of the session. The Home Practice after treatment aims to assure continued progress with LE use after the intervention program is completed. The LE-MAL Log will be administered in all sessions to assess quality of movement of the affected leg, level of assistance needed to perform daily activities, and level of confidence.
  Participants will be assessed pre-, post-intervention, 3 and 6 months after the intervention.
Arm/Group | Treadmill Training +Transfer Package (TT+TP) | Treadmill Training (TT)
Number analyzed (Participants) | 8 | 6
score on a scale
  Total score Pre-treatment | 6.3 (1.11) | 6.4 (1.11)
  Total score Post-treatment | 7.3 (1.02) | 7.2 (0.82)
  Total score 3 months Follow up | 7.4 (1.16) | 7.5 (0.65)
  Total score 6 months Follow up | 7.8 (1.10) | 7.5 (0.74)
Statistical Analysis 1: Comparison: Treadmill Training +Transfer Package (TT+TP) vs Treadmill Training (TT); Considering the small sample size, a descriptive analysis of means and standard deviations was conducted comparing scores obtained on pre-, post-treatment, at the 3- and 6-month follow up assessments visits; Test type: Superiority — Since this is a descriptive analysis, no power calculation was conducted; A descriptive analysis of means and standard deviations was conducted comparing scores obtained on pre-, post-treatment, at the 3- and 6-month follow up assessments visits. Changes in the scores obtained on all time points compared to pre-treatment were also identified

2. Primary Outcome: Berg Balance Scale - Balance Assessment
Description: It is a valid and reliable tool to assess balance control in both static and dynamic activities with people with different health conditions. The Berg includes 14 balance tasks, each one scored from 0 (inability to perform or need for maximum assistance) to 4 (able to perform the task without difficulty or independently). The total score range from 0-56 and a score lower than 44 represents high risk of falling.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Training +Transfer Package (TT+TP) | Treadmill Training (TT)
Number analyzed (Participants) | 8 | 6
score on a scale
  Pre-treatment | 44.8 (5.52) | 47.5 (3.69)
  Post-treatment | 46.4 (5.17) | 50.2 (3.62)
  3 months follow-up | 46.3 (4.2) | 50.0 (3.51)
  6 months follow-up | 44.8 (5.76) | 48.8 (3.62)
Statistical Analysis 1: Comparison: Treadmill Training +Transfer Package (TT+TP) vs Treadmill Training (TT); [analysis description as in outcome 1, analysis 1]; Test type: Other — Since this is a descriptive analysis, no power calculation was conducted; A descriptive analysis of means and standard deviations was conducted comparing scores obtained on pre-, post-treatment, at the 3- and 6-month follow up assessment visits. Changes in the scores obtained on all time points compared to pre-treatment were also identified

3. Primary Outcome: 10 Meters Walk Test - Walking Speed Assessment
Description: It is a gait speed measurement, which is an easy and reliable assessment of locomotion. In this assessment, the individual is asked to walk 10 meter, with or without an assistive decide, and the speed is calculated according to the time the individual takes from the beginning to the end of the 10 meter trail. During the self-selected speed, the individual is asked to walk at his/her/their normal speed, as if the person is walking at home. On the fast speed, the individual is asked to speed up and walk fast as he/she/they can, but not running.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Treadmill Training +Transfer Package (TT+TP) | Treadmill Training (TT)
Number analyzed (Participants) | 8 | 6
meters/second
  Self-selected speed pre-treatment | 0.42 (0.16) | 0.46 (0.21)
  Self-selected speed post-treatment | 0.46 (0.19) | 0.50 (0.20)
  Self-selected speed 3-month follow-up | 0.53 (0.23) | 0.59 (0.26)
  Self-selected speed 6-month follow-up | 0.52 (0.25) | 0.65 (0.28)
  Fast speed pre-treatment | 0.56 (0.27) | 0.59 (0.26)
  Fast speed post-treatment | 0.60 (0.29) | 0.64 (0.30)
  Fast speed 3-month follow-up | 0.70 (0.34) | 0.76 (0.34)
  Fast speed 6-month follow-up | 0.66 (0.35) | 0.74 (0.32)
Statistical Analysis 1: Comparison: Treadmill Training +Transfer Package (TT+TP) vs Treadmill Training (TT); [analysis description as in outcome 1, analysis 1]; Test type: Other — A descriptive analysis of means and standard deviations was conducted comparing scores obtained on pre-, post-treatment, at the 3- and 6-month follow up assessments visits; [other analysis details as in outcome 2, analysis 1]

4. Secondary Outcome: 5-times-sit-to-stand - Functional Strength Assessment
Description: Functional strength assessment tool. In this assessment, the individual is asked to stand up and sit on a chair 5 times and the time spend to perform the task is recorded. A performance time longer than 12 seconds is considered abnormal.
Time Frame: as for outcome 1
Population: COVID has impacted the duration of the treatment that changed from 8 to 6 weeks. Two individuals from TT group were not able to complete this test in one or more of the assessments visits, therefore, for this test, just 4 out of 6 individuals were included in the analysis. Four individuals of the TT+TP group were not able to complete this test in one or more of the assessments visits, therefore, for this test, just 4 out of 8 individuals were included in the analysis.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Treadmill Training +Transfer Package (TT+TP) | Treadmill Training (TT)
Number analyzed (Participants) | 4 | 4
Seconds
  Pre-treatment | 18.3 (2.59) | 20.3 (4.2)
  Post-treatment | 17.2 (1.70) | 18.0 (3.74)
  3-month Follow-up | 17.0 (1.80) | 17.0 (4.79)
  6-month Follow-up | 14.7 (1.31) | 14.7 (3.88)
Statistical Analysis 1: Comparison: Treadmill Training +Transfer Package (TT+TP) vs Treadmill Training (TT); Test type: Other — A descriptive analysis of means and standard deviations was conducted comparing scores obtained on pre-, post-treatment, at the 3- and 6-month follow up assessments visits. Changes in scores post-treatment vs. pre-treatment, and 3 and 6-month follow up vs. post-treatment were calculated; [other analysis details as in outcome 2, analysis 1]

5. Secondary Outcome: 6-minutes Walking Test - Energy Expenditure Assessment.
Description: It is a tool to assess energy expenditure and endurance during walking. The total distance in meters that the individual walked in a 6 minutes period is recorded.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Treadmill Training +Transfer Package (TT+TP) | Treadmill Training (TT)
Number analyzed (Participants) | 8 | 6
Meters
  Pre-treatment | 147.1 (70.05) | 168.2 (72.67)
  Post-treatment | 170.5 (71.89) | 184.5 (81.05)
  3-month Follow-up | 191.2 (77.88) | 212.4 (92.27)
  6-month Follow-up | 185.9 (82.48) | 223.8 (107.57)
Statistical Analysis 1: Comparison: Treadmill Training +Transfer Package (TT+TP) vs Treadmill Training (TT); Test type: Other — [test comment as in outcome 4, analysis 1]; [other analysis details as in outcome 2, analysis 1]

6. Secondary Outcome: Fear of Falling Avoidance Questionnaire - Avoidance Behavior Assessment
Description: In this assessment, the individuals are asked about activities that they avoid due to their fear of falling. It is a questionnaire that identifies how the fear of falling has affected the performance of 14 activities scored from 0 to 4 where 0 means "I completely disagree that I avoid this activity because I am afraid of falling", and 4 means "I completely agree that I avoid this activity because I am afraid of falling". The total score ranges from 0 to 56 where higher scores indicate higher number of activities avoided due to their fear of falling.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treadmill Training +Transfer Package (TT+TP) | Treadmill Training (TT)
Number analyzed (Participants) | 8 | 6
units on a scale
  Pre-treatment | 16.3 (9.87) | 14.0 (9.00)
  Post-treatment | 16.0 (8.87) | 12.8 (6.77)
  3-month Follow up | 16.1 (5.58) | 16.3 (5.85)
  6-month Follow up | 14.1 (6.23) | 13.2 (4.56)
Statistical Analysis 1: Comparison: Treadmill Training +Transfer Package (TT+TP) vs Treadmill Training (TT); Test type: Other — [test comment as in outcome 4, analysis 1]; [other analysis details as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and collected throughout the duration of the intervention. COVID affected the duration of the program, which changed from the initial 8 weeks of duration to 6 weeks. Thus, adverse events of each participant were monitored and collected during 6 weeks.
Description: The definition of the adverse events from clnicaltrials.gov was followed in this study.
Groups:
- Treadmill Training +Transfer Package (TT+TP): The TT+TP group received 18 sessions (3x week for 6 weeks) of robotic treadmill gait training in a robotic device called KineAssist. In combination with the gait training, participants in this group also received a group of behavioral strategies called the "Transfer Package" (TP). Each intervention session will last 1.5h, 1h for the gait training and 30 minutes dedicated for the transfer package. As part of the TP Participants signed the behavioral contract to achieve safety while engaging in activities, increase use of the paretic leg in daily activities, and increase coordination of both legs. A list of activities to be performed outside the clinical setting, the Home Skill Assignment, was developed for each day of the week during the treatment period and given to the participants at the end of the session. The Home Practice after treatment aims to assure continued progress with LE use after the intervention program is completed. The LE-MAL Log was administered in all sessions to assess quality of movement of the affected leg, level of assistance needed to perform daily activities, and level of confidence.
  Participants will be assessed pre-, post-intervention, 3 and 6 months after the end of the intervention.
- Treadmill Training (TT): The TT group received 18 sessions (3x week for 6 weeks) of robotic treadmill gait training in a robotic device called KineAssist. Participants in this group walked doe 30 minutes, in different speeds, and different resistance (strength training). The treadmill training was identical to the experimental group, but no element of the Transfer Package was delivered. In combination with the gait training, participants in this group will receive handouts with a list of exercises suggested by the American Stroke Association. Participants will be assessed pre-, post-intervention, 3 and 6 months after the end of the intervention.
Arm/Group | Treadmill Training +Transfer Package (TT+TP) | Treadmill Training (TT)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/7
Other Adverse Events (participants affected / at risk) | 0/12 | 0/7

LIMITATIONS AND CAVEATS:
This study was affected by the COVID pandemic in multiple ways. The initial sample of 24 had to change to a minimum of 18 due to time constraints, leading us to a smaller sample that did not allow us to follow the planned statistical analysis. Due to institutional restrictions, the duration of the training changed to 6 weeks, instead of the planned 8 weeks. The recruitment was also impacted since all eligible participants were considered high risk of severe symptoms if exposed to the virus.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT04546217/Prot_SAP_001.pdf